CLINICAL TRIAL: NCT00975975
Title: Basiliximab #2: In-Vivo Activated T-Cell Depletion to Prevent GVHD After Nonmyeloablative Allotransplantation for the Treatment of Blood Cancer
Brief Title: Basiliximab #2: In-Vivo Activated T-Cell Depletion to Prevent Graft-Versus_Host Disease (GVHD) After Nonmyeloablative Allotransplantation for the Treatment of Blood Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0908-04; IUCRO-0256
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2016-02-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphocytic Leukemia; Chronic Myelogenous Leukemia; Chronic Lymphocytic Leukemia; Myelodysplasia; Non-Hodgkin's Lymphoma; Hodgkin's Disease; Multiple Myeloma; Myelofibrosis; Anemia, Aplastic; Hemoglobinuria, Paroxysmal
Keywords: Paroxysmal nocturnal hemoglobinuria; severe aplastic anemia; Mantle cell
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Anemia, Refractory, with Excess of Blasts; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Primary Myelofibrosis; Anemia, Aplastic; Hemoglobinuria, Paroxysmal | interventions — Basiliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Basiliximab (Experimental): Basiliximab will be given by IV on Day +7 post transplant for recipients of matched unrelated cells. Basiliximab will be given by IV on Day +9 post transplant for recipients of matched related cells.
  Interventions: Drug: Basiliximab

INTERVENTIONS:
Drug: Basiliximab — Basiliximab given 1 time on Day +7 or Day +9.
  Other Names: Simulect

SUMMARY:
The purpose of this study is to compare the effects (good and bad) of the medication basiliximab in combination with cyclosporine (investigational therapy) for the prevention of a complication of bone marrow transplantation known as graft-versus-host disease (GVHD). GVHD is a complication in which the cells of the transplanted bone marrow react against organs and tissues.

DETAILED DESCRIPTION:
This study is for patients with a blood condition or myelodysplasia (bone marrow disease) which has either not responded to treatment or is not treatable by conventional/routine medical treatments. Bone marrow transplantation is a medical treatment that involves giving high doses of chemotherapy followed by the transplantation of the blood-forming and immune cells from a relative or from a "matched" unrelated person through the National Marrow Donor Program, in an attempt to cure disease in the recipient (the person receiving the donated cells). Nonmyeloablative (bone-marrow preservation) bone marrow transplantation is a relatively new technique in which lower than usual doses of chemotherapy are given before transplantation, in hopes of reducing adverse side effects of the chemotherapy in transplant patients. Nonmyeloablative bone marrow transplantation has several advantages which doctors have determined are beneficial for this condition.

This research is being done because the complication of graft-versus-host disease can be bad for a person and there is no completely safe and effective way to prevent this complication. We know that cyclosporine helps but would like to know if the addition of basiliximab, given with cyclosporine, will decrease the incidence and/or severity of graft-versus-host disease after a transplant known as nonmyeloablative or "mini" transplant.

ELIGIBILITY:
Inclusion Criteria:

* Acute myelogenous leukemia:

  * Second or subsequent remission; patient over 18 yrs of age.
  * Relapsed after autologous HC transplant, over 18 years of age.
  * First remission, Philadelphia chromosome + over age 18.
  * Secondary AML, in first or subsequent remissions.
* Acute lymphocytic leukemia:

  * Philadelphia chromosome + over the age of 50, first or subsequent remission.
  * Relapse following Autologous HC transplantation, ages over 50.
  * Second or subsequent remission over the age of 50
* Chronic myelogenous leukemia:

  * First or second chronic phase over the age of 18.
  * Accelerated phase over the age of 18.
  * Must have failed or been intolerant to a standard tyrosine kinase inhibitor.
* Chronic lymphocytic leukemia:

  * Failed nucleoside-based therapy, ages >18.
* Myelodysplasia:

  * All-risk categories, age greater than 18.
* Non-Hodgkin's Lymphoma, less than 76 years of age

  * Relapsed diffuse aggressive NHL (intermediate and high grade) that fails to achieve CR or PR to conventional salvage chemotherapy.
  * Aggressive NHL includes diffuse large B cell lymphoma, diffuse mixed small and large cell lymphoma, follicular lymphoma for grade 3 (follicular large cell lymphoma), T or B cell lymphoblastic lymphoma, diffuse small noncleaved (Burkett's or Burkett-like ) lymphoma, mantle cell lymphoma, peripheral T cell lymphoma, anaplastic large cell lymphoma, and other diffuse aggressive lymphomas that are not otherwise classifiable
  * Aggressive NHL that has relapsed following autologous HCT. Patients that respond to additional treatment for post-transplant relapse are eligible.
  * Aggressive NHL that does not achieve CR or PR with primary chemotherapy (i.e., primary induction failure).
  * Low-grade lymphoma refractory to standard therapy, including the following:

    1. small cell lymphocytic lymphoma,
    2. follicular lymphoma of grades 1 and 2 (follicular small cleaved and follicular mixed small and large cell lymphoma)
    3. marginal cell lymphoma, splenic lymphoma),
    4. lymphoplasmacytic lymphoma and
    5. other lymphomas not otherwise classifiable.
* Patients with low-grade lymphoma must have experienced progressive disease after receiving three or more of the following regimens:

  * alkylator-based therapy (cyclophosphamide/ vincristine/ prednisone) chlorambucil, monoclonal antibody based therapy (e.g., rituximab, Campath-1H, radiolabelled CD20+ antibodies);
  * nucleoside analog-based therapy (e.g., fludarabine, cladribine).)
* Patients with marginal zone lymphoma or gastric MALT type associated with Helicobacter pylori infection must have progressed after receiving appropriate antibiotic therapy as well as three or more regimens as described above
* Mantle cell, ages 18-75.
* Hodgkin's Disease, ages 18-75.

  * Relapsed or refractory disease after autologous transplant.
* Multiple Myeloma, ages 18-75

  * Recurrent disease after two medical therapies
  * Relapse following autologous transplant
* Myelofibrosis, age greater than 18 years
* Severe aplastic anemia (refractory to immunosuppressive therapy); age greater than 18 years

  * Patients with aplastic anemia must have marrow cellularity ≤ 10% plus 2 of the following:

    1. Absolute granulocyte count <500/mm3
    2. Corrected reticulocyte count <1%
    3. Untransfused platelet count <20,000/mm3 on at least 2 occasions
    4. Hemoglobin <9 g/dL (adults) or < 8 g/dL (children) on at least 2 occasions
* Paroxysmal nocturnal hemoglobinuria; age greater than 18 years.

  * Renal function: creatinine greater than 2.5
* Donor Requirement:

  * Must have a fully HLA-matched (10 of 10 Antigen matched) related or unrelated donor, eighteen years of age or older, who is capable of undergoing GCSF mobilization and apheresis

Exclusion Criteria:

* Active CNS disease (the presence of leukemic blasts in the CSF)
* Pregnancy or breast-feeding.
* Inability to give informed consent.
* AST, ALT, total bilirubin >3x upper limit of normal.
* Creatinine > 2 or creatinine clearance < 50mL/hr. If patient has a creatinine of > 2 or creatinine clearance < 50mL/hr and it is due to the disease process then the patient will not be excluded based on this.
* Fractional shortening by echocardiogram not within normal limits per institution or LVEF of < 40 %.
* Pulmonary function: DLCO not within institutional normal limits or DLCO less than 45% of normal predicted, corrected for anemia
* Prior allogeneic transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-09; Primary Completion 2012-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Nelson, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This protocol has 17 patients. The study was stopped prior to 20 due to the meeting of a stopping rule of 5 or more deaths within the first 15 patients. An additional patient was enrolled after the stopping rule was met. This patient was followed for safety/AE but is not included in the analysis of the efficacy measures, as recommended by the IRB.
Groups:
- Overall: Patients administered 40 mg of basiliximab as a single intravenous dose on day +7, +8, or +9 following infusion of allogeneic peripheral blood hematopoietic cells
Period: Overall Study
Arm/Group | Overall
Started | 17
Completed | 11
Not Completed | 6
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Arm/Group | Overall
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (7.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Grade 3-4 Acute GVHD Rate
Description: The percent of patients where a patient experienced a Grade 3 or 4 acute GVHD
Time Frame: Transplant (Day 0) up to 1 year
Population: All patients enrolled and received treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Overall
Number analyzed (Participants) | 17
percentage of participants | 29.4 [10.3 to 56.0]

2. Secondary Outcome: Time to Neutrophil Engraftment
Description: Time to neutrophil engraftment will be analyzed by the Kaplan-Meier method. The time to engraftment of neutrophils is defined as the time from day 0 to the date of the first of three consecutive days after transplantation during which the absolute neutrophils count (ANC) is at least 0.5 x109/l. Patients who did not have neutrophil engraftment before death will be censored at the date of death. The median and 95% confidence intervals will be provided.
Time Frame: Transplant (Day 0) up to 1 year
Population: All patients enrolled and received treatment, excluding the patient who entered after the stopping rule was met.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Overall
Number analyzed (Participants) | 16
days | 13.5 [10.0 to 14.0]

3. Secondary Outcome: Time to Platelet Engraftment
Description: Time to platelet engraftment will be analyzed by the Kaplan-Meier method. The time to engraftment of platelets is defined as the time from day 0 to the first of seven consecutive days after transplantation during which the platelet count is at least 20 x109/l without transfusion support. Patients who did not have platelet engraftment before death will be censored at the date of death. The median and 95% confidence intervals will be provided.
Time Frame: Transplant (Day 0) up to 1 year
Population: All patients enrolled and received treatment, excluding the patient who entered after the stopping rule was met.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Overall
Number analyzed (Participants) | 16
days | 12.0 [8.0 to 18.0]

ADVERSE EVENTS:
Time Frame: From transplant until the end of the study, for up to 2 years
Arm/Group | Overall
Serious Adverse Events (participants affected / at risk) | 7/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=17)
CARDIAC ARRHYTHMIA - OTHER (Cardiac disorders) | 1
CONDUCTION ABNORMALITY/ATRIOVENTRICULAR HEART BLOCK - ASYSTOLE (Cardiac disorders) | 1
DIARRHEA (Gastrointestinal disorders) | 2
GASTROINTESTINAL - OTHER (Gastrointestinal disorders) | 1
PAIN - ABDOMEN NOS (Gastrointestinal disorders) | 2
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 1
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 2
ALLERGIC REACTION/HYPERSENSITIVITY (INCLUDING DRUG FEVER) (Immune system disorders) | 1
INFECTION (DOCUMENTED CLINICALLY OR MICROBIOLOGICALLY) WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E (Infections and infestations) | 1
INFECTION - OTHER (Infections and infestations) | 4
INFECTION WITH UNKNOWN ANC - BLOOD (Infections and infestations) | 2
INFECTION WITH UNKNOWN ANC - UPPER AIRWAY NOS (Infections and infestations) | 1
THROMBOSIS/EMBOLISM (VASCULAR ACCESS-RELATED) (Injury, poisoning and procedural complications) | 1
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 1
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 1
CREATININE (Investigations) | 2
PLATELETS (Investigations) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1
PAIN - HEAD/HEADACHE (Nervous system disorders) | 1
ADULT RESPIRATORY DISTRESS SYNDROME (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2
PULMONARY/UPPER RESPIRATORY - OTHER (SPECIFY, __) (Respiratory, thoracic and mediastinal disorders) | 1
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=17)
HEMOLYSIS (E.G., IMMUNE HEMOLYTIC ANEMIA, DRUG-RELATED HEMOLYSIS) (Blood and lymphatic system disorders) | 3
LYMPHATICS - OTHER (Blood and lymphatic system disorders) | 1
PALPITATIONS (Blood and lymphatic system disorders) | 1
PETECHIAE/PURPURA (HEMORRHAGE/BLEEDING INTO SKIN OR MUCOSA) (Blood and lymphatic system disorders) | 1
CARDIAC ARRHYTHMIA - OTHER (Cardiac disorders) | 3
CARDIAC GENERAL - OTHER (Cardiac disorders) | 1
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA - ATRIAL FIBRILLATION (Cardiac disorders) | 2
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA - ATRIAL TACHYCARDIA/PAROXYSMAL ATRIAL TACHYCARDIA (Cardiac disorders) | 1
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA - SINUS BRADYCARDIA (Cardiac disorders) | 3
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA - SINUS TACHYCARDIA (Cardiac disorders) | 5
VENTRICULAR ARRHYTHMIA - PVCS (Cardiac disorders) | 1
AUDITORY/EAR - OTHER (Ear and labyrinth disorders) | 2
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1
DRY EYE SYNDROME (Eye disorders) | 1
OCULAR/VISUAL - OTHER (Eye disorders) | 1
VISION-BLURRED VISION (Eye disorders) | 2
VITREOUS HEMORRHAGE (Eye disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 4
DIARRHEA (Gastrointestinal disorders) | 14
DISTENSION/BLOATING, ABDOMINAL (Gastrointestinal disorders) | 3
DYSPHAGIA (DIFFICULTY SWALLOWING) (Gastrointestinal disorders) | 3
ESOPHAGITIS (Gastrointestinal disorders) | 1
FLATULENCE (Gastrointestinal disorders) | 1
GASTROINTESTINAL - OTHER (Gastrointestinal disorders) | 2
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 2
HEMORRHOIDS (Gastrointestinal disorders) | 3
ILEUS, GI (FUNCTIONAL OBSTRUCTION OF BOWEL, I.E., NEUROCONSTIPATION) (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 11
PAIN - ABDOMEN NOS (Gastrointestinal disorders) | 6
PAIN - DENTAL/TEETH/PERIDONTAL (Gastrointestinal disorders) | 2
ULCER, GI - ESOPHAGUS (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 10
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 3
FEBRILE NEUTROPENIA (FEVER OF UNKNOWN ORIGIN WITHOUT CLINICALLY OR MICROBIOLOGICALLY DOCUMENTED INFE (General disorders) | 8
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 14
HOT FLASHES/FLUSHES (General disorders) | 1
HYPOTHERMIA (General disorders) | 1
PAIN - OTHER (General disorders) | 8
RIGORS/CHILLS (General disorders) | 4
SWEATING (DIAPHORESIS) (General disorders) | 3
ASCITES (NON-MALIGNANT) (Hepatobiliary disorders) | 2
BILIRUBIN (HYPERBILIRUBINEMIA) (Hepatobiliary disorders) | 14
ALLERGIC REACTION/HYPERSENSITIVITY (INCLUDING DRUG FEVER) (Immune system disorders) | 2
ALLERGIC RHINITIS (INCLUDING SNEEZING, NASAL STUFFINESS, POSTNASAL DRIP) (Immune system disorders) | 2
INFECTION (DOCUMENTED CLINICALLY OR MICROBIOLOGICALLY) WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E (Infections and infestations) | 1
INFECTION - OTHER (Infections and infestations) | 14
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - BLOOD (Infections and infestations) | 1
INFECTION WITH UNKNOWN ANC - BLOOD (Infections and infestations) | 2
INFECTION WITH UNKNOWN ANC - COLON (Infections and infestations) | 1
INFECTION WITH UNKNOWN ANC - LUNG (PNEUMONIA) (Infections and infestations) | 2
INFECTION WITH UNKNOWN ANC - ORAL CAVITY-GUMS (GINGIVITIS) (Infections and infestations) | 1
INFECTION WITH UNKNOWN ANC - SINUS (Infections and infestations) | 2
INFECTION WITH UNKNOWN ANC - SKIN (CELLULITIS) (Infections and infestations) | 1
INFECTION WITH UNKNOWN ANC - UPPER AIRWAY NOS (Infections and infestations) | 6
INFECTION WITH UNKNOWN ANC - URINARY TRACT NOS (Infections and infestations) | 5
THROMBOSIS/EMBOLISM (VASCULAR ACCESS-RELATED) (Injury, poisoning and procedural complications) | 1
ALKALINE PHOSPHATASE (Investigations) | 12
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 14
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 14
CREATININE (Investigations) | 14
IRON OVERLOAD (Investigations) | 1
MUCOSITIS/STOMATITIS (CLINICAL EXAM) - ORAL CAVITY (Investigations) | 5
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Metabolism and nutrition disorders) | 7
ANOREXIA (Metabolism and nutrition disorders) | 2
CALCIUM, SERUM-HIGH (HYPERCALCEMIA) (Metabolism and nutrition disorders) | 1
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Metabolism and nutrition disorders) | 4
DEHYDRATION (Metabolism and nutrition disorders) | 1
EDEMA: HEAD AND NECK (Metabolism and nutrition disorders) | 2
EDEMA: LIMB (Metabolism and nutrition disorders) | 14
EDEMA: TRUNK/GENITAL (Metabolism and nutrition disorders) | 1
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Metabolism and nutrition disorders) | 9
GLUCOSE, SERUM-LOW (HYPOGLYCEMIA) (Metabolism and nutrition disorders) | 1
MAGNESIUM, SERUM-LOW (HYPOMAGNESEMIA) (Metabolism and nutrition disorders) | 6
PHOSPHATE, SERUM-LOW (HYPOPHOSPHATEMIA) (Metabolism and nutrition disorders) | 3
POTASSIUM, SERUM-HIGH (HYPERKALEMIA) (Metabolism and nutrition disorders) | 1
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Metabolism and nutrition disorders) | 4
SODIUM, SERUM-LOW (HYPONATREMIA) (Metabolism and nutrition disorders) | 4
ARTHRITIS (NON-SEPTIC) (Musculoskeletal and connective tissue disorders) | 1
JOINT-FUNCTION (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL/SOFT TISSUE - OTHER (Musculoskeletal and connective tissue disorders) | 3
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1
PAIN - BACK (Musculoskeletal and connective tissue disorders) | 4
PAIN - BONE (Musculoskeletal and connective tissue disorders) | 3
PAIN - EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 6
PAIN - JOINT (Musculoskeletal and connective tissue disorders) | 4
PAIN - MUSCLE (Musculoskeletal and connective tissue disorders) | 2
PAIN - NECK (Musculoskeletal and connective tissue disorders) | 2
CONFUSION (Nervous system disorders) | 3
CONSTIPATION (Nervous system disorders) | 1
DIZZINESS (Nervous system disorders) | 4
ENCEPHALOPATHY (Nervous system disorders) | 1
INSOMNIA (Nervous system disorders) | 3
NEUROLOGY - OTHER (Nervous system disorders) | 3
NEUROPATHY: MOTOR (Nervous system disorders) | 1
NEUROPATHY: SENSORY (Nervous system disorders) | 2
PAIN - HEAD/HEADACHE (Nervous system disorders) | 7
SEIZURE (Nervous system disorders) | 1
TREMOR (Nervous system disorders) | 7
MOOD ALTERATION - ANXIETY (Psychiatric disorders) | 1
MOOD ALTERATION - DEPRESSION (Psychiatric disorders) | 4
PSYCHOSIS (HALLUCINATIONS/DELUSIONS) (Psychiatric disorders) | 2
BLADDER SPASMS (Renal and urinary disorders) | 1
PAIN - BLADDER (Renal and urinary disorders) | 2
RENAL FAILURE (Renal and urinary disorders) | 2
RENAL/GENITOURINARY - OTHER (Renal and urinary disorders) | 3
URINE COLOR CHANGE (Renal and urinary disorders) | 1
SEXUAL/REPRODUCTIVE FUNCTION - OTHER (Reproductive system and breast disorders) | 1
VAGINAL DRYNESS (Reproductive system and breast disorders) | 1
APNEA (Respiratory, thoracic and mediastinal disorders) | 1
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1
BRONCHOSPASM, WHEEZING (Respiratory, thoracic and mediastinal disorders) | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 9
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 12
HICCOUGHS (HICCUPS, SINGULTUS) (Respiratory, thoracic and mediastinal disorders) | 3
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 9
PAIN - CHEST WALL (Respiratory, thoracic and mediastinal disorders) | 3
PAIN - CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 1
PAIN - THROAT/PHARYNX/LARYNX (Respiratory, thoracic and mediastinal disorders) | 3
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 5
PULMONARY/UPPER RESPIRATORY - OTHER (Respiratory, thoracic and mediastinal disorders) | 3
DERMATOLOGY/SKIN - OTHER (Skin and subcutaneous tissue disorders) | 3
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 2
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 5
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 11
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 3
SKIN BREAKDOWN/DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 2
HEMORRHAGE, GI - LOWER GI NOS (Vascular disorders) | 3
HEMORRHAGE, GI - VARICES (RECTAL) (Vascular disorders) | 1
HEMORRHAGE, GU - BLADDER (Vascular disorders) | 1
HEMORRHAGE, GU - URINARY NOS (Vascular disorders) | 2
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY - NOSE (Vascular disorders) | 2
HEMORRHAGE/BLEEDING - OTHER (Vascular disorders) | 3
HYPERTENSION (Vascular disorders) | 5
HYPOTENSION (Vascular disorders) | 5
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes